CLINICAL TRIAL: NCT04853511
Title: Biological Interconnection Between Stress-associated Neurobiological Activity and Atherosclerotic Plaque Instability: A Prospective Cohort Study With OCT-FLIM Dual-modal Intravascular Imaging and Serial 18F-FDG-PET/CT Assessment
Brief Title: Comprehensive Assessment of Interconnection Between Brain Emotional Activity and Coronary Plaque Instability
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Jin Won Kim, Principal Investigator, Korea University Guro Hospital
Other Study IDs: SRFC-IT1501-05_a
Record Dates: First submitted 2021-04-05; First posted 2021-04-21 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Atherosclerosis, Coronary; Emotional Stress; Inflammation; Hematopoiesis; Atherosclerosis Coronary Artery With Angina Pectoris; Atheroma; Heart; Atherosclerosis; Acute Coronary Syndrome
Keywords: PET-CT; Fluorescence lifetime imaging; Optical coherence tomography; High-risk plaque; Amygdalar activity; Arterial Inflammation; Hematopoietic activity; Biochemical imaging
MeSH Terms: conditions — Coronary Artery Disease; Stress, Psychological; Inflammation; Atherosclerosis; Acute Coronary Syndrome; Arteritis | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OCT-FLIM dual modal intravascular imaging with serial 18F-FDG-PET/CT assessment: Group of patients undergoing PCI with comprehensive assessment of coronary plaque with OCT-FLIM dual modal intravascular imaging followed by serial 18F-FDG-PET/CT imaging
  Interventions: Device: OCT-FLIM (optical coherence tomography-fluorescence life time)

INTERVENTIONS:
Device: OCT-FLIM (optical coherence tomography-fluorescence life time) — comprehensive assessment of coronary plaque with OCT-FLIM dual modal intravascular catheter imaging followed by serial 18F-FDG-PET/CT imaging
  Other Names: 18F-FDG-PET/CT (positron emission tomography-computed tomography)

SUMMARY:
Emotional stress is associated with future cardiovascular events. However, the biological interconnection between brain emotional neural activity and acute plaque instability is not fully understood. Optical coherence tomography-Fluorescence Lifetime (OCT-FLIM) dual modal intravascular imaging is a novel technique that enables comprehensive assessment of structural and biochemical characteristics of coronary atheroma and estimates the level of plaque instability. 18F-fluorodeoxyglucose-positron emission tomography/computed tomography (18F-FDG-PET/CT) enables simultaneous estimation of multi-system activities including emotional stress, arterial inflammation, and hematopoiesis. The present study aims to prospectively investigate mechanistic linkage between coronary plaque instability, stress-associated neurobiological activity, and macrophage hematopoiesis using OCT-FLIM and 18F-FDG PET/CT imaging assessment.

DETAILED DESCRIPTION:
Thirty two patients with multivessel coronary artery disease (including both stable angina and acute coronary syndrome), who have at least one severe obstructive lesion (>70% diameter stenosis) that is considered suitable for percutaneous coronary intervention (PCI), will be included in the study.

Structural/biochemical characteristics of coronary culprit plaque (with or without mild to moderate stenotic non-culprit plaque) will be assessed comprehensively using OCT-FLIM dual modal intravascular imaging.

After coronary revascularization with PCI, subjects will undergo serial 18F-FDG-PET/CT molecular imaging at baseline admission and 6-month follow-up to measure PET signal activities at target tissues including amygdala, carotid artery, aorta, bone marrow, and spleen.

Correlation between OCT-FLIM parameters and baseline PET signals will be assessed to provide insight into the mechanistic linkage between multi-system metabolic activities and coronary plaque instability. Serial PET/CT imaging after 6 month will enable estimation of natural course of multi-system PET signal activities according to different levels of coronary plaque instability.

ELIGIBILITY:
Inclusion Criteria:

* Age: greater than 20, less than 75
* Patients with severe coronary atherosclerosis (diameter stenosis >70%) requiring coronary revascularization
* Reference vessel diameter: between 2.5 and 4.0 mm
* Obtained informed consent from voluntary participants before study enrollment

Exclusion Criteria:

* Complex coronary lesion (ostial lesion, unprotected left main lesion, chronic total occlusion, grafted vessels, etc)
* Reference vessel diameter: less than 2.5 mm, greater than 4.0 mm
* Coronary lesion with heavy calcification
* Hemodynamic instability during coronary intervention
* Contraindication to antithrombotic therapy
* Chronic renal insufficiency (Serum creatinine >2.0mg/dL)
* Severe liver dysfunction (aspartate transaminase or alanine transferase > 5 times of upper normal limit)
* Pregnancy or potential pregnancy
* Life expectancy less than 1 year
* Patient refused to sign the informed consent at enrollment

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are planned to undergo percutaneous coronary intervention with utilization of OCT-FLIM dual modal intravascular imaging for culprit plaque assessment and stent optimization. After PCI, subjects will undergo serial 18F-FDG-PET/CT molecular imaging at baseline and 6-month follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Baseline amygdalar activity (Stress-associated neurobiological activity) | Baseline (within index admission)
  Amygdalar target-to-background ratio (TBR) = Amygdalar standardized uptake value (SUV) / Temporal lobe SUV

SECONDARY OUTCOMES:
Baseline carotid inflammation (arterial atherosclerotic inflammation) | Baseline (within index admission)
  Carotid TBR = Carotid SUV / Jugular vein SUV
Baseline aortic inflammation (arterial atherosclerotic inflammation) | Baseline (within index admission)
  Aorta TBR = Aorta SUV / Jugular vein SUV
Baseline bone marrow hematopoiesis (hematopoietic activity) | Baseline (within index admission)
  Bone marrow TBR = Bone marrow SUV / Jugular vein SUV
Baseline splenic hematopoiesis (hematopoietic activity) | Baseline (within index admission)
  Spleen TBR = Spleen SUV / Jugular vein SUV
Coronary plaque composition estimated by OCT-FLIM | Baseline (day 1)
  Fluorescence Lifetime values that predicts detailed coronary plaque composition

OTHER OUTCOMES:
Follow-up amygdalar activity (Stress-associated neurobiological activity) | 6-month follow-up
  Amygdalar TBR = Amygdalar SUV / Temporal lobe SUV
Follow-up carotid inflammation (arterial atherosclerotic inflammation) | 6-month follow-up
  Carotid TBR = Carotid SUV / Jugular vein SUV
Follow-up aortic inflammation (arterial atherosclerotic inflammation) | 6-month follow-up
  Aorta TBR = Aorta SUV / Jugular vein SUV
Follow-up bone marrow hematopoiesis (hematopoietic activity) | 6-month follow-up
  Bone marrow TBR = Bone marrow SUV / Jugular vein SUV
Follow-up splenic hematopoiesis (hematopoietic activity) | 6-month follow-up
  Spleen TBR = Spleen SUV / Jugular vein SUV

CONTACTS AND LOCATIONS:
Overall Officials: Jin Won Kim, MD, PhD, Principal Investigator — Korea University Guro Hospital; Dong Oh Kang, MD, PhD, Study Director — Korea University Guro Hospital; Sun Won Kim, MD, PhD, Study Director — Korea University; Hongki Yoo, PhD, Study Director — Korea Advanced Institute of Science and Technology
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Due to patient confidentiality, individual participant data (IPD) will not be shared to other researchers.

REFERENCES:
- [Background] Tawakol A, Ishai A, Takx RA, Figueroa AL, Ali A, Kaiser Y, Truong QA, Solomon CJ, Calcagno C, Mani V, Tang CY, Mulder WJ, Murrough JW, Hoffmann U, Nahrendorf M, Shin LM, Fayad ZA, Pitman RK. Relation between resting amygdalar activity and cardiovascular events: a longitudinal and cohort study. Lancet. 2017 Feb 25;389(10071):834-845. doi: 10.1016/S0140-6736(16)31714-7. Epub 2017 Jan 12. PMID 28088338
- [Background] Lee MW, Song JW, Kang WJ, Nam HS, Kim TS, Kim S, Oh WY, Kim JW, Yoo H. Comprehensive intravascular imaging of atherosclerotic plaque in vivo using optical coherence tomography and fluorescence lifetime imaging. Sci Rep. 2018 Sep 28;8(1):14561. doi: 10.1038/s41598-018-32951-9. PMID 30267024
- [Background] Kim S, Yoo H, Kim JW. Long Journey of Intravascular Imaging: What and How to Look at the Atheroma in Coronary Artery. JACC Cardiovasc Imaging. 2021 Sep;14(9):1843-1845. doi: 10.1016/j.jcmg.2020.11.015. Epub 2020 Dec 16. No abstract available. PMID 33341412